CLINICAL TRIAL: NCT00789321
Title: A Randomized Clinical Trial to Evaluate the Effects of Multiple Doses of Amlodipine 10 mg on Pedal Edema Measurements in Middle-Aged and Elderly Healthy Subjects and Patient With Hypertension
Brief Title: A Study to Evaluate Methodologies for Measuring Swelling of the Leg and Ankle (MK-0000-106)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0000-106; 2008_580
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Results first posted 2010-07-08 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): amlodipine
  Interventions: Drug: Comparator: amlodipine besylate
- 2 (Placebo Comparator): Placebo to amlodipine
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: Comparator: amlodipine besylate — Two 5 mg tablets amlodipine daily for 6 weeks.
  Arms: 1
Drug: Comparator: Placebo — Two 5 mg tablets placebo to amlodipine daily for 6 weeks
  Arms: 2

SUMMARY:
This study will evaluate methodologies for measuring pedal edema associated with calcium channel blockers in middle-aged and elderly subjects and patients with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patient does not have hypertension or has Stage I or II hypertension and is taking < 3 anti-hypertension medications
* Patient is willing to discontinue all anti-hypertensive medications during study
* Patient is willing to refrain from drinking alcohol for 24 hours prior to each study visit and is willing to limit intake at other times during the study to 2 drinks per day
* Patient agrees to avoid caffeine for 24 hours prior to each study visit. At other times during study, daily caffeine intake should not exceed 4 cups of coffee (or equivalent)
* Patient will avoid strenuous physical activity during study
* Patient is a nonsmoker or has not smoked for the last 3 months

Exclusion Criteria:

* Patient has metal implants in the leg or artificial limbs
* Patient has had a lower limb amputation, malformation, alterations in leg muscles, or a history of musculoskeletal disease
* Patient has used oral contraceptive pills or hormone replacement therapy within 3 months of screening
* Patient has a history of stroke or seizures
* Patient has a history of cancer, except that which was treated at least 10 years prior to screening and shows no evidence of recurrence

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2008-07; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Schoeller DA, Alon A, Manekas D, Mixson LA, Lasseter KC, Noonan GP, Bolognese JA, Heymsfield SB, Beals CR, Nunes I. Segmental bioimpedance for measuring amlodipine-induced pedal edema: a placebo-controlled study. Clin Ther. 2012 Mar;34(3):580-92. doi: 10.1016/j.clinthera.2012.01.018. Epub 2012 Mar 3. PMID 22385927

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited across 3 Phase I clinical research units in the US. Participants participated from July 2008 to March 2009.
Pre-assignment Details: Participants taking anti-hypertensive medications at screening were required to washout of this therapy before randomization and remain off the therapy during the study. Participants were eligible if systolic blood pressure (BP) was ≥120 to <180 mm Hg and diastolic BP was ≥80 to <110 mm Hg at screening (or after 2-4 weeks of washout, if applicable)
Groups:
- Amlodipine 10 Milligrams: Participants who were randomized to treatment with amlodipine 10 mg once daily for 6 weeks
- Placebo: Participants who were randomized to treatment with placebo once daily for 6 weeks
Period: Overall Study
Arm/Group | Amlodipine 10 Milligrams | Placebo
Started | 24 | 23
Completed | 24 | 22
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amlodipine 10 Milligrams | Placebo | Total
Number analyzed (Participants) | 24 | 23 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (5.6) | 59.6 (6.2) | 59.0 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 11 | 12 | 23
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.2 (2.9) | 29.0 (2.7) | 28.6 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Segmental Bioimpedance Measurements at 10 Kilohertz (KHz) at Week 2
Description: Segmental biomimpedance was measured using a multifrequency analyzer (ImpediMed SFB7). The device was used to measure impedance (measured in Ohms) of a small current traveling between leads placed at the ankle and knee. Least Squares Mean Difference from Baseline in impedance is the primary endpoint.
Time Frame: Baseline and 2 weeks
Population: All patients treated with segmental bioimpedance measurements at baseline and 2 weeks - one patient in the placebo group was not included (dropped out of study due to viral infection prior to Week 2).
Measure: Least Squares Mean (Standard Deviation); unit: Ohms
Arm/Group | Amlodipine 10 Milligrams | Placebo
Number analyzed (Participants) | 24 | 22
Ohms | -7.9 (20.7) | 3.8 (17.0)
Statistical Analysis 1: Comparison: Amlodipine 10 Milligrams vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA; Change from baseline in systolic blood pressure included as covariate; Least Squares Mean = -11.7, 90% CI [-18.1 to -5.4]

2. Secondary Outcome: Change From Baseline in Foot Volume by Water Displacement (Weight of Water Displaced) at Week 2
Description: Least Squares Mean Difference from Baseline
Time Frame: Baseline and 2 weeks
Population: All patients treated with water displacement measurements at baseline and 2 weeks - one patient in the placebo group was not included (dropped out of study due to viral infection prior to Week 2) - two patients in the amlodipine group were excluded due to technical/procedural errors.
Measure: Least Squares Mean (Standard Deviation); unit: Grams
Arm/Group | Amlodipine 10 Milligrams | Placebo
Number analyzed (Participants) | 22 | 22
Grams | 44.8 (64.8) | 5.8 (53.2)
Statistical Analysis 1: Comparison: Amlodipine 10 Milligrams vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA; Change from baseline in systolic blood pressure included as covariate; Least Squares Mean = 39.0, 95% CI [17.9 to 60.1]

ADVERSE EVENTS:
Arm/Group | Amlodipine 10 Milligrams | Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 17/24 | 16/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amlodipine 10 Milligrams (N=24) | Placebo (N=23)
Palpitations (Cardiac disorders) | 1 | 0
Myodesopsia (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Feeling Hot (General disorders) | 1 | 0
Inflammation (General disorders) | 0 | 1
Oedema Peripheral (General disorders) | 12 | 9
Pyrexia (General disorders) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Viral Infection (Infections and infestations) | 0 | 1
Accidental Overdose (Injury, poisoning and procedural complications) | 3 | 2
Arthropod Bite (Injury, poisoning and procedural complications) | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Tension Headache (Nervous system disorders) | 1 | 2
Euphoric Mood (Psychiatric disorders) | 1 | 0
Polyuria (Renal and urinary disorders) | 1 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.